CLINICAL TRIAL: NCT03398551
Title: Machine Learning From Fetal Flow Waveforms to Predict Adverse Perinatal Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Universitat Pompeu Fabra (Other)
Responsible Party: Principal Investigator, Zahra Hoodbhoy, Dr Zahra Hoodbhoy, Aga Khan University
Other Study IDs: 4872-Ped-ERC-17
Record Dates: First submitted 2018-01-06; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Perinatal Mortality; Neonatal Morbidities
Keywords: pregnancy; machine learning; fetal Doppler echocardiography
MeSH Terms: conditions — Perinatal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to get a proof of concept for using a computational model of fetal haemodynamics, combined with machine learning based on Doppler patterns of the fetal cardiovascular, cerebral and placental flows, to identify those at increased risk of adverse perinatal outcomes such as stillbirth, perinatal mortality and other neonatal morbidities.

We will also compare the sensitivity and specificity of UmbiFlow device with the machine learning model in predicting adverse perinatal outcomes

DETAILED DESCRIPTION:
Pakistan is one of the countries where stillbirth rate (43/1000 total births) and neonatal mortality rate (55/1000 live births) are among the highest in the world. The figures for perinatal mortality remained unchanged between Pakistan Demographic and Health Survey (PDHS) 1990-91 and PDHS 2012-13. It is hence important to evaluate new techniques to identify high-risk pregnant women who can then subsequently receive personalized care to improve perinatal outcomes. Fetal blood flow waveforms assessed via Doppler ultrasound to indicate wellbeing of the fetus have been in practice for nearly four decades. Abnormal blood flow patterns in the fetal circulation detected by Doppler ultrasound may indicate poor fetal prognosis. These tracings will then be incorporated in a computational model and combined with machine learning, will be used to predict adverse perinatal outcomes.

This will be a prospective one group cohort study for a period of twelve months which will be based in Ibrahim Hyderi, a peri-urban settlement of approximately 70,000 on the south east of Karachi. The sample size for this study has been calculated based on the outcomes of the pregnancy and was estimated to be 525 pregnant women.

Recruitment - Household surveillance will be done by community health workers (CHWs) in the catchment area in a sequential manner to identify pregnant women. Eligible women between 22-34 weeks of gestation on last menstrual period (LMP) will then be explained regarding the purpose of the study and invited for an ultrasound scan.

First and enrollment visit - The first visit window for the ultrasound scan will be between 22-26 weeks of gestation. This window is selected because pregnancies at risk may be better identified and also visualization of fetal cardiac flow is possible. Based on the rigorous surveillance, we anticipate that most women will be in this window. The following information will be collected:

* Socio-demographic information
* Medical history, including exposure to tobacco, gravidity, parity, past obstetric history (including number of miscarriages, stillbirths or neonatal deaths) and comorbid conditions (pre-eclampsia, diabetes mellitus)
* Maternal anthropometry (height, weight and mid-upper arm circumference)
* Maternal blood pressure
* Hemoglobin of the mother
* Symphysiofundal height will be measured
* Standard obstetric Doppler evaluation including the four primary ultrasound measures of fetal growth-head circumference, biparietal diameter, abdominal circumference, and femur length is routinely performed for all pregnant women presenting at the center. These parameters will be used to estimate fetal weight (automatically calculated by the machine).
* Focused Fetal Doppler Echocardiography - These would include transabdominal measurements of the Doppler velocity of the umbilical artery, the middle cerebral artery (MCA), ductus arteriosus, fetal aortic isthmus (AoI) and left and right ventricular outflow tracts
* UmbiFlow - Umbilical artery continuous wave Doppler image will also be obtained on these women. The device will generate graphs for the flow pattern and calculate the resistance index for the flow.

Second visit - The second visit window of ultrasound scan will be between 30-34 weeks of gestation. This will be applicable for all women who have had their first scan during 22-26 weeks of gestation as well as newly enrolled women during 30-34 weeks of gestational age. Cardiotocography (CTG) will be performed for all recruited women during the second visit followed by the Doppler examination. The same procedures as described in the first visit will be done.

Follow up - We will obtain contact information (phone number) from all enrolled women. A trained research midwife will be responsible for making phone calls, as well as performing household visits at pre-specified intervals for immediate and early identification of the pregnancy outcome. A team of CHWs will perform home visits to the baby at post-natal day 1 and 6 and questions related to delayed cry, neonatal sepsis and hospital course (if any) will be collected and the weight and length of the baby will be recorded.

Verbal autopsy - The VA team will visit the family after the grieving period (at least 14 days after the death). VA will be performed using a structured tool (http://www.who.int/healthinfo/statistics/WHO_VA_2012_RC1_Instrument.pdf ).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman coming to the ultrasound clinic between 22-34 weeks of gestation.
* Written informed consent
* Resident of the study area

Exclusion Criteria:

* Multiple gestation
* Known congenital anomaly in the fetus or newborn
* Refusal for the ultrasound
* Poor echocardiographic images for Doppler acquisition

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — This study will recruit pregnant women only.
Study Population: Pregnant women between 22-34 weeks who reside in Ibrahim Hyderi Goth which is a peri-urban settlement of approximately 70,000 on the south east of Karachi. It is one of the seven union councils in Bin Qasim town which has a population of one million.
Sampling Method: Non-Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Stillbirth | At birth
  Baby born with no signs of life at or after 28 weeks of gestation
Early neonatal mortality | Within the first 7 days of life
  Death of a baby within the first 7 days of life

SECONDARY OUTCOMES:
IUGR | At birth
  Fetal weight that is below the 10th percentile for gestational age as determined through an ultrasound
Prematurity | At birth
  Birth of a fetus at < 37 weeks of gestation
Birth asphyxia | At birth
  Delayed cry after at least 1 minute of life
Neonatal sepsis | Within the first 7 days of life
  Any 1 of the following danger signs: fever > 38 of < 35.5 C, convulsions, lethargy, poor feeding, chest in drawing and tachypnea (respiratory rate > 60/min)
Low Birth Weight | At birth
  Birth weight < 2.5 kg

IPD SHARING:
Plan to Share IPD: Undecided